CLINICAL TRIAL: NCT02734654
Title: Pulmonary Remote Preconditioning by Ischemia-reperfusion in Lung Lobectomy. A Study on the Prevention of Oxidative Stress
Brief Title: Limb RIPC in Patients Undergoing Lung Lobectomy. Study of Oxidative Lung Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, José García de la Asunción, MD, PhD, Instituto de Salud Carlos III
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI070836
Record Dates: First submitted 2016-03-28; First posted 2016-04-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Acute Lung Injury
Keywords: oxidative stress; lung lobectomy
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): patients do not receive remote preconditioning prior to lung lobectomy
- RIPC group (Experimental): patients receive remote preconditioning prior to lung lobectomy
  Interventions: Procedure: remote ischemic preconditioning (RIPC)

INTERVENTIONS:
Procedure: remote ischemic preconditioning (RIPC) — Remote ischemic preconditioning: The limb RIPC was applied after the induction of anaesthesia and consisted of 3 cycles: 5 min of ischemia by a cuff-inflator on a thigh and inflated to 200 mmHg, followed by 5 min deflated. The control group had during the same time a deflated cuff on a thigh.
  Arms: RIPC group

SUMMARY:
Background: In patients undergoing lung lobectomy, lung collapse and re-expansion after resection is associated to severe oxidative lung injury. The researchers hypothesized that remote ischemic preconditioning (RIPC) could reduce oxidative lung injury and improve the oxygenation parameters.

Methods: We designed a single-centre, randomized, prospective and double-blind study, conducted in fifty-three patients with non-small cell lung cancer undergoing elective lung lobectomy.

Fifty-three patients were randomly assigned to 2 groups: 26 patients received limb RIPC (3 cycles: 5 min ischemia/5 min reperfusion induced by an ischemia cuff applied on the thigh) and 27 controls.

Time course of oxidative stress marker levels was simultaneously studied in exhaled breath condensate (EBC) and blood at four specific time points: T0, pre-operatively; T1, during operated lung collapse and one-lung ventilation (OLV); T2, immediately after resuming two-lung ventilation (TLV); T3, 120 min after resuming TLV.

EBC 8-isoprostane was the primary outcome. Secondary outcomes included PaO2/FiO2, other pulmonary oxygenation variables, other oxidative markers (NO2-+NO3-, H2O2) and pH.

DETAILED DESCRIPTION:
In patients with non-small-cell lung carcinoma (NSCLC), the surgical resection remains the primary and preferred approach to the treatment of stage I-II NSCLC. Despite advances in surgical techniques, these patients have a risk of development a severe lung injury, because during lobectomy the operated lung is completely collapsed and hypoperfused. This hypoperfusion is due in part to a reactive hypoxic pulmonary vasoconstriction in response to alveolar hypoxia, which optimizes gas exchange. Hypoxic or ischemic tissues increase the reactive oxygen species (ROS) production in mitochondria respiratory chain, because the respiratory cytochromes become redox-reduced allowing them to directly transfer electrons to O2 producing large amount of superoxide anions, which contributes to more vasoconstriction. The primary site of ROS production during hypoxia appears to be complex III, and paradoxical increase of ROS production during hypoxia may be explained by an effect of O2 within mitochondria inner membrane on the ubisemiquinone radical in complex III. Thus, patients undergoing lobar resection suffer a relative lung ischemia-hypoxia during the collapse, followed by expansion-reperfusion injury attributed to the production of ROS. Acute lung injury (ALI) and postoperative adult respiratory distress syndrome (ARDS) after major thoracic surgery remains the leading cause of death from pulmonary surgery. Because to date few studies have assessed this subject in detail, we have showed recently also an increase of oxidative stress damage during lung lobectomy, associated to a direct correlation of lung collapse time with oxidative stress marker levels in exhaled breath condensate and blood.

Remote ischemic preconditioning (RIPC) has emerged as a procedure for different organs protection against acute ischemia/reperfusion injury as is shown by different clinical trials. Although most studies have been conducted in patients undergoing coronary artery by-pass grafting and valvular heart surgery, also were observed protective effect in other organs as kidneys, intestine and others. RIPC is an innate and powerful mechanism where a tissue or organ is exposed to a transient episode of ischemia-reperfusion and then confer a global resistance to subsequent episodes of ischemia in remote organs. However the potential mechanism through which RIPC works is unclear. The signal transfer to organs is through humoral, neuronal and systemic communications, which activate specific receptors, intracellular kinases and mitochondrial function. Recently has been reported that limb RIPC attenuates intestinal and pulmonary injury after abdominal aortic aneurysm repair and also after pulmonary resection, where they found significant decreases in serum malondialdehyde in treated group with RIPC.

EBC collection is non-invasive method for obtain samples from the lower respiratory tract, which contains large number of biomarkers including isoprostanes, nitrogen oxides and hydrogen peroxide. The isoprostanes are a family of products from arachidonic acid produced by the non-enzymatic action of ROS. Increased blood level of 8-isoprostane is considered a reliable index of lipid peroxidation in vivo due to its chemical stability. NO. and superoxide anion (O2.-) react to form ONOO-, which is a powerful oxidant. Nitrites (NO2-) and nitrates (NO3-) are end products of nitric oxide (NO.) and peroxynitrite anion (ONOO-) metabolism and present in the epithelial lining fluid of the respiratory tract. Hydrogen peroxide (H2O2) is a ROS and volatile molecule produced from conversion of superoxide anion (O2.-) to H2O2 by superoxide dismutase and released from inflammatory and epithelial cells of respiratory system.

The aim of this study is to investigate whether RIPC would reduce the oxidative lung injury in cancer patients undergoing lung lobectomy. The primary outcome of this study was compare 8-isoprostene and others oxidative marker levels in EBC and blood between patients receiving RIPC and control patients. Also to evaluate whether there is a correlation between OLV duration and oxidative stress marker levels in EBC and blood.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer patients (clinical stage I-II NSCLC)
* elective lung lobectomy
* patients were randomized and prospectively studied in a single centre
* all patients were ASA physical status I-II category
* pregnants

Exclusion Criteria:

* previous radiotherapy-chemotherapy
* previous thorax surgery
* PaO2 <60 mmHg
* FEV1 <50%
* cardiac disease (NYHA II-IV)
* active infections and temperature >37.5 ºC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-11; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Time course of 8-isoprostane levels in exhaled breath condensate during and after lung lobectomy | Approximately 4 hours: after anesthesia (T0), during lung lobectomy (T1, T2) and 2 hours after lung lobectomy (T3)
  levels of 8-isoprostane in exhaled breath condensate were measured during lung lobectomy (T0: after anesthesia induction; T1: before two lung ventilation; T3: after two lung ventilation) and 2 hours after lobectomy in critical care unit (T3).

SECONDARY OUTCOMES:
Time course of PO2/FiO2 ratio in arterial blood gas during and after lung lobectomy | during lung lobectomy (T0, T1, T2) and 24 hours after lung lobectomy in the critical care unit (T3, T4, T5)
  PO2/FiO2 ratio in arterial blood gas during lung lobectomy and during 24 hours in critical care unit

CONTACTS AND LOCATIONS:
Overall Officials: José García de la Asunción, MD, PhD, Principal Investigator — Instituto de Investigador Sanitaria, INCLIVA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-de-la-Asuncion J, Garcia-Del-Olmo E, Galan G, Guijarro R, Marti F, Badenes R, Perez-Griera J, Duca A, Delgado C, Carbonell J, Belda J. Glutathione oxidation correlates with one-lung ventilation time and PO2/FiO2 ratio during pulmonary lobectomy. Redox Rep. 2016 Sep;21(5):219-26. doi: 10.1080/13510002.2015.1101890. Epub 2016 Jan 21. PMID 26795138
- [Background] Misthos P, Katsaragakis S, Theodorou D, Milingos N, Skottis I. The degree of oxidative stress is associated with major adverse effects after lung resection: a prospective study. Eur J Cardiothorac Surg. 2006 Apr;29(4):591-5. doi: 10.1016/j.ejcts.2005.12.027. Epub 2006 Feb 14. PMID 16476542
- [Background] Horvath I, Hunt J, Barnes PJ, Alving K, Antczak A, Baraldi E, Becher G, van Beurden WJ, Corradi M, Dekhuijzen R, Dweik RA, Dwyer T, Effros R, Erzurum S, Gaston B, Gessner C, Greening A, Ho LP, Hohlfeld J, Jobsis Q, Laskowski D, Loukides S, Marlin D, Montuschi P, Olin AC, Redington AE, Reinhold P, van Rensen EL, Rubinstein I, Silkoff P, Toren K, Vass G, Vogelberg C, Wirtz H; ATS/ERS Task Force on Exhaled Breath Condensate. Exhaled breath condensate: methodological recommendations and unresolved questions. Eur Respir J. 2005 Sep;26(3):523-48. doi: 10.1183/09031936.05.00029705. PMID 16135737
- [Background] Przyklenk K, Whittaker P. Remote ischemic preconditioning: current knowledge, unresolved questions, and future priorities. J Cardiovasc Pharmacol Ther. 2011 Sep-Dec;16(3-4):255-9. doi: 10.1177/1074248411409040. PMID 21821525
- [Result] Garcia-de-la-Asuncion J, Garcia-del-Olmo E, Perez-Griera J, Marti F, Galan G, Morcillo A, Wins R, Guijarro R, Arnau A, Sarria B, Garcia-Raimundo M, Belda J. Oxidative lung injury correlates with one-lung ventilation time during pulmonary lobectomy: a study of exhaled breath condensate and blood. Eur J Cardiothorac Surg. 2015 Sep;48(3):e37-44. doi: 10.1093/ejcts/ezv207. Epub 2015 Jun 18. PMID 26088589